CLINICAL TRIAL: NCT04056858
Title: Identification and Investigation of a Gene Involved in Monogenic Forms of Goldenhar Syndrome.
Brief Title: Study of a Candidate Gene Involved in Goldenhar Syndrome.
Acronym: GOLDGEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHU BX 2012/11
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Goldenhar Syndrome; Oculoauriculovertebral Dysplasia
Keywords: array-CGH; exome sequencing
MeSH Terms: conditions — Goldenhar Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The informed consent of the patients has already been gathered during the genetic consultation prior to any molecular analysis.
  The samples received are:
  - 2 tubes of blood on EDTA or 1 aliquot of DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to identify of the first gene involved in the Goldenhar syndrome in a cohort of 120 affected patients.

DETAILED DESCRIPTION:
Goldenhar syndrome belongs to the heterogeneous spectrum of oculoauriculovertebral dysplasia. Several chromosomal abnormalities have been described associated with this spectrum, and furthermore mutations in different genes of development cause abnormalities of the jaw or facial asymmetries in human or mouse. To date, no gene has been identified as formally involved in the genesis of the OAVS, despite evidence of familial cases, mostly with autosomal dominant inheritance.

The aim of this study is to identify of the first gene involved in the Goldenhar syndrome in a cohort of 120 affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Spectrum of oculoauriculovertebral dysplasia minimal features include unilateral microtia and hemifacial microsomia

Exclusion Criteria:

* Absence of minimal spectrum of oculoauriculovertebral dysplasia features, molecular anomaly identified, other diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of 120 patients affected with Goldenhar/spectrum of oculoauriculovertebral dysplasia , whose phenotype is finely characterized, and that were analyzed using an oligonucleotide array-CGH pangenomic approach
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2012-09-29 (Actual); Primary Completion 2014-01-08 (Actual); Study Completion 2014-01-08 (Actual)

PRIMARY OUTCOMES:
presence of sequence variation | At the screening
  Identification of the first gene involved in Goldenhar syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ROORYCK THAMBO, Dr, Principal Investigator — Bordeaux Universitu Hospital

IPD SHARING:
Plan to Share IPD: No